CLINICAL TRIAL: NCT04334720
Title: PET/MRI Study on the Effects of Psychosocial on Fat and Muscle Metabolism for Malignant Tumor Patient After Comprehensive Treatment.
Brief Title: PET/MRI Study on Changes of Fat and Muscle Metabolism.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Fat & Muscle -No.1
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Brown Fat and Muscle Metabolic; Differential Diagnosis
Keywords: Psychological; Comprehensive treatment; Positron emission computed tomography/Magnetic resonance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Observation group of positive F&M: The baseline PET/MR scan was performed before comprehensive treatment, and the contrast scan was performed after treatment and the sequence and protocol was consistent. Get psychological assessment before and after treatment and the time interval shall not exceed half a year
  Interventions: Other: Comprehensive treatment of tumor
- Observation group of no abnormal changes in F&M: The baseline PET/MR scan was performed before comprehensive treatment, and the contrast scan was performed after treatment and the sequence and protocol was consistent. Get psychological assessment before and after treatment and the time interval shall not exceed half a year
  Interventions: Other: Comprehensive treatment of tumor
- The control group: Corresponding to the observation group, the time, sequence and protocol were consistent

INTERVENTIONS:
Other: Comprehensive treatment of tumor — According to the pathologic types and TNM stage of tumor，specialists chose one or more of the interventions in surgery, radiotherapy, chemotherapy, targeted therapy and immunotherapy.
  Groups: Observation group of no abnormal changes in F&M; Observation group of positive F&M

SUMMARY:
False positives for Brown Fat & Muscle（F&M） always affect the evaluation of metabolic disease treatment. Recently, using PET/CT，international journals such as Journal of Nuclear Medicine reported that the amount of active brown fat was correlated with renal creatinine clearance and subject to regulation by atrial natriuretic peptide in addition to association of season and temperature. At present，studies based on PET/CT have shown that elimination of the above factors, brown fat(even muscle) will still appear false positive metabolism in tumor patients. In view of the basis of Positron emission computed tomography/Magnetic resonance (PET/MRI) brain function research，our team speculate that it may be related to psychological or cortex metabolism. And there is a lack of studies on the correlation between the psychosocial，cortex structure and metabolism. Therefore, it suggests that，combination of structure and metabolism，PET/MRI will play a role in studying the effects of psychological on F&M false-positive metabolism in malignant patients. In this project, the investigators intend to observe the changes of F&M metabolism with psychological and cortex metabolism after comprehensive treatment in malignant patient by combining PET/MRI. The relationship between F&M metabolism and psychological will be deeply analyzed to provide scientific basis for the development of the differential diagnosis and assessment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of malignant tumor
* Have not yet been receiving comprehensive treatment and should begin within one month
* Fasting glucose of diabetic patients is controlled below 11.1 mmol/L.

Inclusion Criteria for Healthy Control Participants:

• Clinical diagnosis of Healthy Control

Exclusion Criteria:

* Fasting glucose ≥11.1mmol/L
* History of endocrine disease (such as chronic glomerulonephritis, Addison's disease)
* Neurological signs and/or history of neurological disease
* Have begun comprehensive treatment
* Presence of magnetically active objects in the body
* Claustrophobia or any other medical condition that would preclude the participant from lying in the PET/MRI scanner for approximately 40 mins.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: patients of the Tangdu hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Change metabolism of glucose of M&F | Baseline, 1 day ( Contrast scanning)
  Glucose metabolic scores will be assessed with visual scale
Change of the glucose metabolism area of M&F | Baseline, 1 day ( Contrast scanning)
  Five different anatomical locations (subphrenic, paravertebral, mediastinal, cervical, supraclavicular) will be assessed with visual.
Change of activated M&F volume | Baseline, 1 day ( Contrast scanning)
  Activated M&F volume before and after comprehensive treatment were evaluated by post-processing software
Change of M&F SUVmax and SUVmean | Baseline, 1 day ( Contrast scanning)
  SUVmax and SUVmean scores will be measured by post-processing software.
Change of anxiety symptoms | Baseline, 1 day ( Contrast scanning)
  Anxiety symptoms scores will be assessed with Hamilton Anxiety Scale.
Change of sleep | Baseline, 1 day ( Contrast scanning)
  Sleep scores will be assessed with Pittsburgh sleep quality index one month before scanning
Change of metabolism of glucose in the M&F | Baseline, 1 day ( Contrast scanning)
  Accumulation of 18F-FDG will be analyzed by treatment-related, psychology-related and intervention-related Positron emission tomography/ Magnetic resonance

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No